CLINICAL TRIAL: NCT01356966
Title: The Role of Neurovascular Dysfunction and Oxidative Stress in the Exercise Intolerance of Renal Failure
Brief Title: Exercise Intolerance in Renal Failure
Acronym: EIRF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeanie Park, Assistant Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00019181; K23HL098744 (NIH)
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — sapropterin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetrahydrobiopterin + Folate (Experimental): Male subjects with hypertension and chronic kidney disease stage 2 or 3 will receive Tetrahydrobiopterin (6R-BH4) 200 mg twice daily and folic acid 1 mg daily
  Interventions: Drug: Tetrahydrobiopterin; Dietary Supplement: Folate
- Placebo + Folate (Placebo Comparator): Male subjects with hypertension and chronic kidney disease stage 2 or 3 will receive 2 placebo pills twice daily and folic acid 1 mg daily
  Interventions: Drug: Placebo; Dietary Supplement: Folate

INTERVENTIONS:
Drug: Tetrahydrobiopterin — Tetrahydrobiopterin (BH4) 200 mg PO BID for 12 weeks
  Other Names: Kuvan
  Arms: Tetrahydrobiopterin + Folate
Drug: Placebo — 2 placebo pills PO BID for12 weeks
  Arms: Placebo + Folate
Dietary Supplement: Folate — Folate 1 mg daily for 12 weeks
  Other Names: Folic Acid

SUMMARY:
Patients with chronic kidney disease have profound exercise intolerance which contributes to an increased risk of cardiovascular disease. The investigators have found that chronic kidney disease patients have an exaggerated increase in blood pressure during certain forms of exercise that could certainly contribute to exercise dysfunction as well as cardiovascular risk. The investigators will test the mechanisms underlying this exaggerated blood pressure response, as well as the potential benefits of short-term tetrahydrobiopterin (BH4) with folic acid on both exercise dysfunction and cardiovascular risk factors in chronic kidney disease. The investigators will test whether short-term treatment with tetrahydrobiopterin (BH4), a cofactor for nitric oxide, together with folic acid improves inflammation, vascular health, and adrenaline levels, both at rest and during exercise in chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease (CKD) stages I, II, and III and do not regularly exercise

  1. CKD Stages I, II, and III will be defined as reduction in estimated glomerular filtration rate (eGFR) to 30-59 cc/minute as calculated by the Modification of Diet in Renal Disease (MDRD) equation, or an eGFR>60 cc/minute with proteinuria greater than 500 mg/g of Creatinine or 500 mg per 24 hours.
* willing and able to cooperate with the protocol
* CKD patients must have stable renal function (no greater than a 20% reduction in eGFR over the prior 3 months)
* controls will be matched for age, gender, race, and hypertensive status.

Exclusion Criteria:

* severe CKD (eGFR<30 cc/minute)
* drug or alcohol abuse
* diabetes
* any serious systemic disease that might influence survival
* severe anemia with hgb level <10 g/dL
* clinical evidence of congestive heart failure or ejection fraction below 35%
* any history of past myocardial infarction or cerebrovascular accident
* symptomatic heart disease determined by electrocardiogram, stress test, and/or history
* treatment with central alpha agonists
* uncontrolled hypertension with BP greater than 160/90 mm Hg
* low blood pressure with BP less than 110/60
* history of nephrolithiasis
* pregnancy or plans to become pregnant
* treatment with vitamin C within the past 3 months
* hepatic enzyme concentrations greater than 2 times the upper limit of normal
* HIV infection
* surgery within the past 3 months
* previous treatment with BH4
* known hypersensitivity to BH4
* any condition that places the participant at high risk of poor adherence or poor follow-up
* patients must be willing to use an acceptable method of contraception if of childbearing age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia

REFERENCES:
- [Derived] Lin AM, Liao P, Millson EC, Quyyumi AA, Park J. Tetrahydrobiopterin ameliorates the exaggerated exercise pressor response in patients with chronic kidney disease: a randomized controlled trial. Am J Physiol Renal Physiol. 2016 May 1;310(10):F1016-25. doi: 10.1152/ajprenal.00527.2015. Epub 2016 Mar 9. PMID 26962106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Atlanta Veterans Affairs (VA) Medical Center from August 2010 to May 2014.
Pre-assignment Details: 42 subjects were withdrawn prior to group assignment. 16 were screen failures, 7 subjects withdrew, and 19 subjects were terminated early.
Groups:
- Tetrahydrobiopterin + Folate: Male subjects with hypertension and chronic kidney disease stage 2 or 3 received Tetrahydrobiopterin (BH4) 200 mg twice daily and folic acid 1 mg daily
- Placebo + Folate: Male subjects with hypertension and chronic kidney disease stage 2 or 3 received 2 placebo pills twice daily and folic acid 1 mg daily
Period: Overall Study
Arm/Group | Tetrahydrobiopterin + Folate | Placebo + Folate
Started | 18 | 14
Completed | 16 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were randomized in the study are included in baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetrahydrobiopterin + Folate | Placebo + Folate | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (1.3) | 55.2 (2.2) | 56.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Muscle Sympathetic Nerve Activity (MSNA)
Time Frame: Baseline, 12 weeks
Population: Two subjects withdrawn from each arm due to adverse events. Additionally, two subjects from the treatment group and one subject from the placebo group were not included in this analysis because an adequate MSNA neurogram was unable to be obtained at the end of the study.
Measure: Mean (Standard Error); unit: bursts/minute
Arm/Group | Tetrahydrobiopterin + Folate | Placebo + Folate
Number analyzed (Participants) | 14 | 11
bursts/minute | -7.5 (2.1) | 3.2 (1.3)

2. Secondary Outcome: Change in Mean Central Augmentation Index (AIx)
Description: The augmentation index (AIx) is a measure of systemic arterial stiffness, and is defined as the ratio of augmentation (Δ P) to central pulse pressure and expressed as percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. The mean AIx for each group was estimated as an average and expressed as a change from baseline to 12 weeks.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: percent
Arm/Group | Tetrahydrobiopterin + Folate | Placebo + Folate
Number analyzed (Participants) | 18 | 14
percent | -5.8 (2.0) | 1.8 (1.7)

3. Secondary Outcome: Change in Heart-rate-corrected Augmentation Index (AIx)
Description: The augmentation index (AIx) is a measure of systemic arterial stiffness, and is defined as the ratio of augmented aortic pressure (Δ P) to central pulse pressure expressed as a percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. Because heart rate (HR) affects AIx, AIx was corrected to a HR of 75 beats per minute (bpm) as follows: HR-corrected AIx = -0.39 x (75 - HR) + AIx. The mean AIx for each group was estimated as an average and expressed as a change from baseline to 12 weeks.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: percent
Arm/Group | Tetrahydrobiopterin + Folate | Placebo + Folate
Number analyzed (Participants) | 18 | 14
percent | -3.2 (2.1) | 1.1 (1.2)

ADVERSE EVENTS:
Arm/Group | Tetrahydrobiopterin + Folate | Placebo + Folate
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 2/18 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetrahydrobiopterin + Folate (N=18) | Placebo + Folate (N=14)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (General disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes